CLINICAL TRIAL: NCT02659384
Title: A Phase II Study of the Anti-PDL1 Antibody Atezolizumab, Bevacizumab and Acetylsalicylic Acid to Investigate Safety and Efficacy of This Combination in Recurrent Platinum-resistant Ovarian, Fallopian Tube or Primary Peritoneal Adenocarcinoma
Brief Title: Anti-programmed Cell Death-1 Ligand 1 (aPDL-1) Antibody Atezolizumab, Bevacizumab and Acetylsalicylic Acid in Recurrent Platinum Resistant Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EORTC-1508; 2015-004601-17 (EudraCT Number)
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; atezolizumab; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bevacizumab (Experimental): Bevacizumab monotherapy treatment in arm 1 will be discontinued upon RECIST documented progression or upon treatment withdrawal, whichever occurs first. Patients will cross-over to the combination of bevacizumab and atezolizumab upon progression as long as they meet cross-over criteria.
  Interventions: Drug: Bevacizumab
- atezolizumab + bevacizumab + placebo (Experimental): The randomized treatment regimen (atezolizumab + bevacizumab + placebo) will be continued until treatment failure or upon treatment withdrawal, whichever occurs first. Patients then go off protocol treatment and further treatment is left to the investigator's decision.
  Interventions: Drug: Bevacizumab; Drug: atezolizumab; Drug: placebo
- atezolizumab + bevacizumab + acetylsalicylic acid (Experimental): The randomized treatment regimen (atezolizumab + bevacizumab + acetylsalicylic acid) will be continued until treatment failure or upon treatment withdrawal, whichever occurs first. Patients then go off protocol treatment and further treatment is left to the investigator's decision.
  Interventions: Drug: Bevacizumab; Drug: atezolizumab; Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
Drug: atezolizumab
  Arms: atezolizumab + bevacizumab + acetylsalicylic acid; atezolizumab + bevacizumab + placebo
Drug: acetylsalicylic acid
  Arms: atezolizumab + bevacizumab + acetylsalicylic acid
Drug: placebo
  Arms: atezolizumab + bevacizumab + placebo

SUMMARY:
This is a randomized phase II study, aimed at evaluating the efficacy (through progression free survival at 6 months) and safety of 5 different treatments involving atezolizumab, bevacizumab and/or acetylsalicylic acid in advanced recurrent platinum-resistant ovarian cancer patients in order to select the optimal treatments for further development in Phase III.

ELIGIBILITY:
Inclusion Criteria:

Recurrent, histologically proven, platinum-resistant, epithelial ovarian, fallopian tube and primary peritoneal cancer in advanced or metastatic stage. Histological diagnosis by image guided biopsy, laparoscopy or laparotomy. Tumors diagnosed on cytology only and borderline tumors are excluded.

At least one lesion accessible to biopsy without putting patient at risk

WHO PS: 0-2 for patients having received no more than two previous lines of therapy. WHO PS: 0-1 for patients having received >2 previous lines of therapy

Prior chemotherapy or bevacizumab:

Any number of platinum-based chemotherapy lines are allowed but a maximum of 2 previous non-platinum containing lines

Prior treatment with bevacizumab or other targeted agents against Vascular Endothelial Growth Factor (VEGF) or VEGF receptor is allowed, but at least 18 weeks must have elapsed since their last administration

Eligible patients with ≤ 2 previous treatment lines must have been previously exposed to bevacizumab or other targeted agents against VEGF or VEGF receptor

Patients may have had prior therapy providing the following conditions are met:

Radiation therapy: wash-out period of 14 days prior to the first study treatment; exception: single fraction radiotherapy with the indication of pain control

Systemic anti-tumor therapy: wash-out period of 21 days prior to the first study treatment

Recovery from any toxic effects of prior therapy to ≤ Grade 1 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.03) except fatigue or alopecia.

Exclusion criteria:

Age <18 years

Life expectancy of < 12 weeks

No adequate hematologic and end organ function

Use of acetylsalicylic acid, NSAIDs or other COX-2 inhibitors that cannot be stopped at baseline and for the whole duration of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) at 6 months assessed by Response Evaluation Criteria in Solid Tumors (RECIST) | 6 months
  Progression Free Survival at 6 months assessed by local investigator

CONTACTS AND LOCATIONS:
Overall Officials: Susana- Banerjee, Study Chair — Royal Marsden Hospital - UK; George Coukos, Study Chair — Centre hospitalier universitaire vaudois, Lausanne
Locations (12):
- France (2):
  - Assistance Publique - Hopitaux de Paris - Hopital Europeen Georges Pompidou, Paris
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
- Netherlands (3):
  - Academisch Medisch Centrum - Universiteit van Amsterdam, Amsterdam
  - Leiden University Medical Centre, Leiden
  - Radboudumc - Radboud University Medical Center Nijmegen, Nijmegen
- Spain (2):
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Badalona
  - Hospital Universitario San Carlos, Madrid
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois - Lausanne, Lausanne
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- United Kingdom (3):
  - Guy's and St Thomas' NHS - Guy s and St Thomas' NHS - Guy's Hospital, London
  - Royal Marsden Hospital - Chelsea, London, London
  - Royal Marsden Hospital - Sutton, Surrey, Sutton

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961